CLINICAL TRIAL: NCT01623349
Title: Phase I Study of the Oral PI3kinase Inhibitor BKM120 or BYL719 and the Oral PARP Inhibitor Olaparib in Patients With Recurrent Triple Negative Breast Cancer or High Grade Serous Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-159
Record Dates: First submitted 2012-06-07; First posted 2012-06-20 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: Recurrent; High Grade; Serous; Triple Negative
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Recurrence | interventions — NVP-BKM120; olaparib; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm BKM (Experimental): BKM120 and Olaparib
  Interventions: Drug: BKM120 and Olaparib
- Arm BYL (Experimental): BYL719 and Olaparib
  Interventions: Drug: BYL719 and Olaparib

INTERVENTIONS:
Drug: BKM120 and Olaparib — Olaparib twice daily (starting dose 50 mg) and BKM120 once daily (starting dose 40 mg). Both drugs are given orally.
  Other Names: Olaparib (NSC 747856); BKM120 (IND 102823)
  Arms: Arm BKM
Drug: BYL719 and Olaparib — Olaparib twice daily (starting dose 100 mg) and BYL719 once daily (starting dose 250 mg). Both drugs are given orally.
  Other Names: Olaparib (NSC 747856); BYL719 (IND 107078)
  Arms: Arm BYL

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational combination of drugs. Phase I studies also try to define the appropriate dose of the investigational combination to use for further studies. "Investigational" means that the combination of these drugs is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved either of these drugs nor the combination of being tested for use in patients, including people with your type of cancer.

BKM120, BYL719 and olaparib are drugs that may stop cancer cells from growing abnormally. These drugs when combined in laboratory experiments with animals, have demonstrated anti-cancer activity. Information from these other research studies suggests that the following agents BKM120, BYL719 and olaparib, may help to shrink tumor cells in the types of cancers being studied in this research study.

In this research study, the investigators are looking for the highest dose that can be given safely and also to see if the combination of BKM120 or BYL719 and olaparib is effective in treating your type of cancer.

DETAILED DESCRIPTION:
During this study, additional tests will be performed on a sample of your original tumor that has been stored in your institutions tissue banks. These tests will be performed on tumor tissue samples from previous biopsies or surgeries for your cancer. The research done on these samples will involve looking at DNA and proteins in your cancer to see if researchers can learn more about your type of cancer and understand how this combination of drugs might work on your tumor. Testing of this sample will not require you to undergo any additional research procedures.

Approximately 2 tablespoons of blood will be collected for research testing. This testing will involve looking at DNA and proteins in your blood to compare them with those seen in your cancer. This will be drawn before you begin taking the study drug.

You may also participate in an optional blood test for the BRCA gene. The BRCA gene test is a blood test that uses DNA analysis to see changes in either one of two breast cancer genes, known as BRCA1 or BRCA2. After having a BRCA gene test performed, you learn whether you carry an inherited BRCA gene mutation. If your blood is tested for the BRCA gene, the results will be reported to your study doctor who will share the results with you and provide information related to your personal risk of breast cancer. Having a BRCA gene mutation is rare, occurring in only about 1 in 1000 people. Inherited BRCA gene mutations are responsible for less than 5 to 10 percent of breast cancers and about 10 to 15 percent of ovarian cancers.

Participants in the dose expansion portion of the study may be asked to have a tumor biopsy done. The dose expansion phase for the combination of BKM120 and Olaparib has been determined. The combination of BYL719 and Olaparib is currently in the dose escalation phase and the dose expansion phase has not been determined. Before and after you begin taking BKM120 (or BYL719) and olaparib, your doctor may also ask you to participate in an optional study where you would have tumor biopsies done.

Participation in the tumor biopsy and blood test for the BRCA gene are optional, and whether you consent or refuse to undergo these additional tests will not affect your participation in the main research study.

Since the investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have high grade serious ovarian cancer or triple negative breast cancer, not everyone who participates in this research study will receive the same dose of the study drug. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

All drugs are in oral form. If you take part in this research study, you will be given a study dosing calendar for each drug for each treatment cycle. Each treatment cycle lasts 4 weeks. BKM120 or BYL719 should be taken once daily in the morning, one hour after a light meal. Olaparib should be taken twice a day continuously, about twelve hours apart. The olaparib morning dose should be taken at the same time as BKM120 or BYL719 one hour after a light meal. The evening dose can also be taken one hour after a light meal or on an empty stomach either 1 hour before or 2 hours after meals. If you vomit either or both medications, record this on your diary and do not take another dose that day.

The investigators will assess your tumor by CT or MRI scan every 8 weeks. During Cycle 1, you will come into the clinic every week, and during cycle 2, you will come into clinic every 2 weeks. For all cycles thereafter, you will come in once every 4 weeks.

During study visits you will undergo some or all of the following: evaluation of performance status, recording of any healthy problems, physical exam including vital signs, list of medications taken since last visit, questionnaire to evaluate anxiety and depression, routine blood tests, research blood tests, Electrocardiogram and optional biopsy.

You will remain in this research study as long as you are benefitting from study treatment. If you are removed from the research study for any reason you may be followed for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent high grade serous ovarian cancer or triple negative breast cancer
* Subjects with recurrent, metastatic triple negative breast cancer must have had at least 1 chemotherapy regimen for metastatic breast cancer or have developed metastatic breast cancer within 1 year of completion of adjuvant chemotherapy
* Prior therapy for high grade serous ovarian cancer subjects must have included a first-line platinum-based regimen
* At least 4 weeks since prior radiation therapy, 3 weeks since prior chemotherapy and 6 weeks if the last regimen included BCNU or mitomycin C
* At least 4 weeks since any small-molecular kinase inhibitors or any other type of investigational agent
* Life expectancy of at least 4 months
* Able to swallow and tolerate oral medications

Exclusion Criteria:

* Evidence of bowel obstruction, abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of study entry
* Current dependency on IV hydration or total parental nutrition
* Diabetes mellitus unless well controlled
* Pregnant or breast feeding
* History of grade 3 or 4 toxicities with previous PI3kinase inhibitor or PARP inhibitor
* Current or active dermatologic diagnoses that would preclude interpretation of skin toxicities of BKM120
* Receiving any medications or substances that are strong inhibitors or inducers of CYP3A4
* History of cardiac dysfunction or disease
* Persistent toxicities (greater than or equal to CTCAE grade 2) caused by previous cancer therapy
* Major surgery within 14 days of starting study treatment
* Evidence of coagulopathy or bleeding diathesis
* History of major depressive episode, bipolar disorder, obsessive/compulsive disorder, schizophrenia, history of suicide attempt or ideation or homicide/homicidal ideation
* CTCAE grade 3 or greater anxiety
* Uncontrolled, intercurrent illness
* Known HIV positive and on combination antiretroviral therapy
* Receiving chronic treatment with steroids or another immunosuppressive agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-09; Primary Completion 2019-05 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Determine MTD and RP2D of the Combination of BKM120 and Olaparib, and the Combination of BYL719 and Olaparib | 2 years
  To determine the maximally tolerated dose (MTD) and recommended phase 2 dose (RP2D) of the combination of BKM120 and olaparib, and the combination of BYL719 and olaparib in patients with recurrent TNBC and HGSC.

SECONDARY OUTCOMES:
Determine the overall Safety and Observed Toxicities of combining BKM120 and Olaparib, and combining BYL719 and Olaparib | 2 years
  To determine the safety and observed toxicities of the combination of BKM120 and olaparib, and the combination of BYL719 and olaparib in this population
Determine Pharmacokinetics of BKM120 and Olaparib, and BYL719 and Olaparib | 2 years
  To measure the drug levels of both BKM120 and olaparib, and both BYL719 and olaparib at different time points after they are started to see if either drug affects the metabolism and levels of the other. PK samples will be drawn in duplicate (one set to be sent to Astrazeneca and the second set to Novartis). BKM120 (or BYL719) and olaparib levels will be performed at the following timepoints:
  1. prior to taking both BKM120 (or BYL719) and olaparib cycle 1, day 1.
  2. Cycle 1, day 8: prior to dosing, 1, 2, 4, and 8 hours post am dosing.
  3. Cycle 1, day 15: prior to dosing, 1, 2, 4, and 8 hours post am dosing.
Determine preliminary activities of these combinations at the MTD and RP2 dose | 2 years
  To determine a preliminary anti-cancer activities of these combinations at the MTD and RP2D dose. Anti-cancer activities of these combinations will be measured by response rate by RECIST 1.1 in patients who have measurable cancer
Exploratory Translational Endpoints | 2 years
  (A) To determine the downstream signaling effects of the PI3-kinase pathway whenboth PI3-kinase and PARP are inhibited.
  (B) To determine BRCA1 immnostaining, BRCA1 promoter hypermethylation and somatic mutations in BRCA1 and BRCA2 in archived formalin fixed paraffin embedded (FFPE) tissue and any new available tissues (pre- or post-treatment biopsies and biopsies or other tumor colelction for clinical care at the time of or following tumor progression)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula A. Matulonis, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Batalini F, Xiong N, Tayob N, Polak M, Eismann J, Cantley LC, Shapiro GI, Adalsteinsson V, Winer EP, Konstantinopoulos PA, D'Andrea A, Swisher EM, Matulonis UA, Wulf GM, Mayer EL. Phase 1b Clinical Trial with Alpelisib plus Olaparib for Patients with Advanced Triple-Negative Breast Cancer. Clin Cancer Res. 2022 Apr 14;28(8):1493-1499. doi: 10.1158/1078-0432.CCR-21-3045. PMID 35149538
- [Derived] Chi P, Qin LX, Camacho N, Kelly CM, D'Angelo SP, Dickson MA, Gounder MM, Keohan ML, Movva S, Nacev BA, Rosenbaum E, Thornton KA, Crago AM, Francis JH, Martindale M, Phelan HT, Biniakewitz MD, Lee CJ, Singer S, Hwang S, Berger MF, Chen Y, Antonescu CR, Tap WD. Phase Ib Trial of the Combination of Imatinib and Binimetinib in Patients with Advanced Gastrointestinal Stromal Tumors. Clin Cancer Res. 2022 Apr 14;28(8):1507-1517. doi: 10.1158/1078-0432.CCR-21-3909. PMID 35110417
- [Derived] Przybytkowski E, Davis T, Hosny A, Eismann J, Matulonis UA, Wulf GM, Nabavi S. An immune-centric exploration of BRCA1 and BRCA2 germline mutation related breast and ovarian cancers. BMC Cancer. 2020 Mar 12;20(1):197. doi: 10.1186/s12885-020-6605-1. PMID 32164626
- [Derived] Konstantinopoulos PA, Barry WT, Birrer M, Westin SN, Cadoo KA, Shapiro GI, Mayer EL, O'Cearbhaill RE, Coleman RL, Kochupurakkal B, Whalen C, Curtis J, Farooq S, Luo W, Eismann J, Buss MK, Aghajanian C, Mills GB, Palakurthi S, Kirschmeier P, Liu J, Cantley LC, Kaufmann SH, Swisher EM, D'Andrea AD, Winer E, Wulf GM, Matulonis UA. Olaparib and alpha-specific PI3K inhibitor alpelisib for patients with epithelial ovarian cancer: a dose-escalation and dose-expansion phase 1b trial. Lancet Oncol. 2019 Apr;20(4):570-580. doi: 10.1016/S1470-2045(18)30905-7. Epub 2019 Mar 14. PMID 30880072